CLINICAL TRIAL: NCT01312311
Title: Phase II Trial of Cisplatin Plus Weekly Docetaxel as the First-line Treatment for Recurrent or Metastatic Nasopharyngeal Cancer
Brief Title: Weekly Docetaxel Plus Cisplatin as the First-line Therapy for Nasopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myung-Ju Ahn / Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-07-005
Record Dates: First submitted 2011-02-21; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Nasopharyngeal Cancer
Keywords: nasopharyngeal cancer; weekly docetaxel; cisplatin
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- weekly docetaxel and cisplatin (Experimental): Docetaxel 35mg/m2 D1 & D8 Cisplatin 70mg/m2 D1 every 3 weeks maxinum 6 cycles
  Interventions: Drug: Docetaxel, Cisplatin

INTERVENTIONS:
Drug: Docetaxel, Cisplatin — Docetaxel 35mg/m2 D1 & D8 Cisplatin 70mg/m2 D1

SUMMARY:
The investigators will evaluate weekly docetaxel plus 3-weekly cisplatin regimen as the first-line therapy for recurrent of metastatic nasophayngeal cancer

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed nasopharyngeal cancer
* chemotherapy or radiotherapy naive (but, including patients completed 6 months before the enrollment)
* ECOG 0-1
* at least one measurable lesion

Exclusion Criteria:

* other cancer
* pregnat
* docetaxel hypersentitivity history
* severe heart or pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 6 months after the enrollment of the last patients

SECONDARY OUTCOMES:
number of patients with adverse events | simultaneously when the analysis of primary endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea